CLINICAL TRIAL: NCT04856631
Title: A Phase Ib/II, Single-arm, Multi-center Clinical Study of Toripalimab Injection (JS001) + Cetuximab in Treatment of Advanced Head and Neck Squamous Cell Cancer
Brief Title: A Study of Toripalimab Injection (JS001) + Cetuximab in Treatment of Advanced Head and Neck Squamous Cell Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-037-Ib/II-HNSCC
Record Dates: First submitted 2021-03-14; First posted 2021-04-23 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Squamous Cell Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Toripalimab Injection (JS001) + Cetuximab
  Interventions: Drug: Toripalimab Injection; Drug: Cetuximab Solution for infusion

INTERVENTIONS:
Drug: Toripalimab Injection — 240mg once per 3 weeks
Drug: Cetuximab Solution for infusion — First infusion 400mg/m2，Subsequent infusions 250mg/m2。once per week

SUMMARY:
This study is a Phase Ib/II, open-label, multicenter clinical trial. Here, the study phase Ib is mainly to evaluate safety of combination regimen of Toripalimab and Cetuximab in treatment of relapsed or metastatic HNSCC failing first-line platinum-based therapy and determine the recommended Phase II dose (RP2D); the study phase II is divided into two cohorts. Cohort A used to evaluate the efficacy and safety of the combination of regimen for relapsed or metastatic HNSCC failing first-line platinum-based regimen containing chemotherapy;cohort B used to evaluate the efficacy and safety of the combination regimen for PD-L1-positive HNSCC that have not received prior systemic therapy for relapsed or metastatic disease.

DETAILED DESCRIPTION:
This study is a Phase Ib/II, open-label, multicenter clinical trial. Here, the study phase Ib is mainly to evaluate safety of combination regimen of Toripalimab and Cetuximab in treatment of relapsed or metastatic HNSCC failing first-line platinum-based therapy and determine the recommended Phase II dose (RP2D); the study phase II is divided into two cohorts. Cohort A used to evaluate the efficacy and safety of the combination of regimen for relapsed or metastatic HNSCC failing first-line platinum-based regimen containing chemotherapy;cohort B used to evaluate the efficacy and safety of the combination regimen for PD-L1-positive HNSCC that have not received prior systemic therapy for relapsed or metastatic disease.

The study consists of the screening period, treatment period, and follow-up period. The screening period is not more than 28 d; after completion of the examinations and assessment in the screening period, eligible subjects enter the investigational therapy period. The subjects will receive the investigational medical product in accordance with the Protocol until radiologically documented progressive disease as judged by the investigator in accordance with RECIST 1.1 criteria, intolerable toxicity, voluntary termination of the treatment or voluntary withdrawal of the informed consent by the subject, or termination of the treatment as judged by the investigator, or until 2 years of JS001 treatment duration (whichever occurs first).

ELIGIBILITY:
Inclusion criteria： 1. Patients voluntarily participate in this study after full informed consent and sign a written informed consent form; 2. Age >=18 to <=75 years at time of consenting; 3. Relapsed or metastatic head and neck squamous cell cancer confirmed histologically or cytologically, and occurred in mouth, oropharynx, laryngopharynx, throat, or paranasal sinus, already being unsuitable to receive local therapy such as surgery or radiotherapy; 4. Phase Ib and Phase II Cohort A:Previously receiving a first-line platinum-based chemotherapy against relapsed or metastatic disease, and developing progressive disease during or after treatment; or receiving platinum-based chemotherapy as neoadjuvant or adjuvant chemotherapy (or chemoradiotherapy), and developing relapse or metastasis within 6 months after end of treatment.

5.Phase II cohort B:

1. No previous systemic treatment for relapsed or metastatic disease. Relapse or metastasis more than 6 months after the end of treatment if previously treated with systemic therapy as part of local treatment.
2. Qualified tumor tissue samples with positive PD-L1 expression (defined as Combined Positive Score (CPS) ≥ 1) tested by the central laboratory are required.

6. All acute toxic reactions from prior antitumor therapy, surgical procedures, or radiotherapy, etc., are relieved to Grades 0-1 (in accordance with NCI-CTCAE version 5.0) or to the level specified in the inclusion/exclusion criteria. Hair loss or pigmentation, or other toxicities that would not result in safety risk to subjects and would not influence compliance, as considered by the investigator, Are ruled out.

7. Previous tumor samples or fresh tumor tissue biopsy samples may be provided.

8 For subjects with oropharyngeal cancer, a prior test report for HPV16 may be provided, or eligible tumor tissue samples are provided to test HPV status.

9. At least one measurable lesion in accordance with RECIST 1.1 assessment criteria;

10 Patients with life expectancy >=12 weeks;

11. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1 point;

12. Good organ function level:

System organ Lab Value

Hematology (no blood transfusion or colony-stimulating factor or other drug correction within 14 days prior to the first study dose)

Neutrophil count ≥1.5×10^9/L

Platelet count ≥100×10^9/L

Hemoglobin ≥90 g/L

Kidney function

Serum creatinine <=1.5 x upper limit of normal (ULN) or Creatinine clearance is calculated with reference to the Cockcroft-Gault formula or the site practices ≥50 mL/min

Hepatic function

total Bilirubin <=1.5 x ULN or<=3 x ULN (patients with known Gilbert's disease)

ALT/AST <=3 x ULN (without liver metastasis) or<=5 x ULN (in case of liver metastases)

Albumin (no infusion of albumin product with 14 days prior to the first dose of the investigational medical product)≥30g/L

Coagulation function

International normalized ratio (INR)

Prothrombin Time (PT)

Activated Partial Thromboplastin Time (aPTT) <=1.5 x ULN

13. Within 72 h prior to the first dose, for women of childbearing age must confirm that the serum pregnancy test is negative and agree to adopt effective contraceptive measures during use of the investigational medical product and for 5 months after last dose. A female of childbearing potential in this Protocol is defined as a sexually mature female who:

1) No hysterectomy or bilateral oophorectomy, 2) Spontaneous menopause does not last for 24 consecutive months (amenorrhea after cancer treatment does not rule out fertility) (i.e., menstruation at any time within the previous 24 consecutive months).

Male patients with partners of childbearing potential must agree to use effective contraception during the use of the investigational medical product and for 5 months after last dose.

Exclusion criteria：

1. Nasopharyngeal cancer or salivary gland cancer confirmed histologically or cytologically, or other non-squamous cell cancer (e.g., adenocarcinoma, sarcoma, or mixed cancer), or metastatic squamous cell cancer with unknown primary site.
2. Patients with necrotic lesion, at risk for major hemorrhage as judged by the investigator.
3. Previously receiving other immune checkpoint inhibitors/drugs acting on immune checkpoint pathway/other drugs acting on T cell costimulation (e.g.: PD-1/PD-L1 antibody or CTLA-4 antibody);
4. Previous treatment of EGFR inhibitor (including radiotherapy sensitization therapy);
5. Diagnosed with other malignancies within 5 years prior to study entry, except for basal cell carcinoma of the skin or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix or carcinoma in situ of the breast that can be cured by local therapy
6. Existing uncontrollable or symptomatic active central nervous system (CNS) metastasis, that may be characterized by clinical symptoms, cerebral edema, spinal cord compression, cancerous meningitis, pia mater disease, and/or progressive growth;

1) Patients with asymptomatic spinal cord compression indicated radiologically may be enrolled, if assessed as stable by the specialist and requiring no treatment presently; 2) Patients who have previously received treatment for CNS metastases, and become stable for >=4 weeks as indicated radiologically in the screening period, and stopped systemic hormone therapy (prednisone in a dose >10 mg/d or an equivalent hormone) for >=4 weeks prior to the first dose of the investigational therapy may be enrolled;

7. Poorly controlled hydrothorax, hydrops abdominis, or pericardial effusion;

8. Existing Grade >=2 (in accordance with NCI-CTCAE 5.0) peripheral neuropathy or hearing loss;

9. Pregnant or breastfeeding female subjects;

10. In the following cases within 6 months prior to the first dose: Myocardial infarction, serious/unstable angina, NYHA Grade >=2 cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, or symptomatic congestive heart failure;

Note: Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be treated with an optimized stable medical regimen at the discretion of the treating physician, with consultation with a cardiologist, as appropriate;

11. Poorly controlled hypertension (systolic blood pressure (BP) >=160 mmHg and/or diastolic blood pressure >=100 mmHg) (based on the mean of >=3 BP readings obtained from >=2 measurements); hypertensive crisis or hypertensive encephalopathy within 6 months prior to the first dose.

12. Patients with known allergy to the investigational medical product or any excipient, or with serious allergic reaction to other monoclonal antibodies;

13. Receiving the following drugs or therapies prior to first dose of investigational medical product :

1. Major surgery within 28 d prior to the first dose of the investigational therapy (tissue biopsy required for diagnosis, and pieripherally inserted central catheter [PICC] or infusion port implantation are permissible).
2. Antitumor therapy (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, cytokine therapy, or biological therapy, etc.) with 28 d prior to the first dose of the investigational medical product;
3. Participation in other intervention studies within 28 d prior to the first dose of the investigational medical product;
4. Treatment with a systemic immunostimulatory drug (including but not limited to interferon or IL-2) within 14 d or 5 half-lives of the investigational medicinal product (whichever is longer) prior to the first dose of the investigational medical product;
5. Treatment of a systemic corticosteroid (> 10 mg/d prednisone or equivalent drug) or other systemic immunosuppressive drugs (including but not limited to Cyclophosphamide, Azathioprine, Methotrexate, Thalidomide and anti-tumor necrosis factor drugs [anti-TNF]) within 14 d prior to the first dose of the investigational therapy;

   o Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are permitted;
   * Patients receiving an acute low-dose systemic immunosuppressive agent (e.g., a single dose of dexamethasone for nausea, or preventive medication prior to administration of Cetuximab ) may be enrolled after discussion with and approval by the medical monitor;
   * Patients who need baseline and follow-up MRI/CT tumor assessment can use steroids prophylaxis if they have previous allergic reactions to intravenous contrast media.
   * Inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for orthostatic hypotension, and low-dose corticosteroids for maintenance treatment of adrenocortical insufficiency are permitted;
6. Treatment of oral or intravenous antibiotic therapy (except preventive use of antibiotics) with 14 d prior to the first dose of the investigational therapy;
7. Vaccination of any live vaccine (e.g., vaccine against infectious diseases, such as influenza vaccine or varicella vaccine, etc.) within 28 d prior to the first dose of the investigational medical product;

14. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, glomerulonephritis;

1. Patients with autoimmune-related hypothyroidism on a stable dose of thyroid hormone replacement are eligible;
2. Patients with type 1 diabetes who are controlled after receiving a stable insulin regimen are eligible for this study;

15. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;

16. Serious infection (NCI-CTCAE Grade >2) within 28 d prior to the first dose of the investigational therapy, e.g., serious pneumonia requiring hospitalization, bacteremia, or infection complications, etc.

17. Active infection, including but not limited to tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, and TB screening according to local medical routine), hepatitis B, hepatitis C or human immunodeficiency virus (HIV antibody positive);

1. Patients who are positive for hepatitis B surface antigen (HBsAg+) and/or hepatitis B core antibody (HBcAb+) are required to undergo hepatitis B virus deoxyribonucleic acid (HBV DNA) test. If HBV DNA copy number is ˂1000 cps/mL or <200 IU/mL, or less than the lower limit of detectable value at the study site, the patients are eligible to participate in this study;
2. Patients who are positive for hepatitis C antibody (HCV Ab+) are required to have an HCV RNA test and are eligible for this study only if they are negative for HCV RNA (defined as below the lower limit of detectable value at the research site);

18. Idiopathic pulmonary fibrosis, drug-induced pneumonia, organized pneumonia (i.e., bronchiolitis obliterans), clinically symptomatic radiation pneumonia or active pneumonia, or those requiring steroid therapy, or other moderate to severe pulmonary diseases influencing seriously pulmonary function.

19. Patients with existing other serious physical or mental disorders or laboratory test abnormalities, or alcoholism or drug abuse, etc., that may increase the risk for participation in the study, influence compliance to the treatment, or interference the study results, or other conditions that are not suitable for participation in the study, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR)evaluated by RECIST 1.1-Phase2 | Up to 2 years
  Evaluate efficacy of the combination therapy in treatment of relapsed or metastatic HNSCC in accordance with the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), as objective response rate (ORR) evaluated
Incidence and severity of adverse event (AE) and serious adverse event (SAE)-Phase1 | Up to 2 years
  Incidence and severity of adverse event (AE) and serious adverse event (SAE) judged in accordance with NCI-CTCAE V5.0; and abnormalities in vital signs, ECG and laboratory tests, etc.

SECONDARY OUTCOMES:
Objective response rate(ORR)evaluated by the investigator-Phase2 | Up to 2 years
  Evaluate efficacy of the combination therapy in treatment of relapsed or metastatic HNSCC in accordance with RECIST 1.1, as objective response rate (ORR) evaluated by the investigator.
Disease control rate（DCR）and Duration of response（DOR）and progression-free survival (PFS).-Phase2 | Up to 2 years
  Evaluate efficacy of the combination therapy in treatment of relapsed or metastatic HNSCC as disease control rate (DCR), duration of response (DOR), and progression-free survival (PFS).
Overall survival（OS） | Up to 2 years
  Evaluate efficacy of the combination therapy in treatment of relapsed or metastatic HNSCC as overall survival (OS) and 1-year OS
Incidence and severity of adverse event (AE) and serious adverse event (SAE) judged in accordance with NCI-CTCAE V5.0 | Up to 2 years
  Incidence and severity of adverse event (AE) and serious adverse event (SAE) judged in accordance with NCI-CTCAE V5.0; and abnormalities in vital signs, ECG and laboratory tests, etc.

OTHER OUTCOMES:
Recommended Phase 2 dose (RP2D)-Phase1 | Up to 2 years
  Recommended Phase 2 dose (RP2D) of the combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China